CLINICAL TRIAL: NCT06820294
Title: Assessing the Clinical Benefits of Whole Genome Sequencing for Children With Neoplasms
Brief Title: Retrospective WGS Study
Status: Enrolling by invitation | Type: Observational
Sponsor: The Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 319310
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Pediatric Cancer; Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All children/young people (up to 21years) diagnosed with neoplastic disorder who have had NHSE WGS: All children and young people (up to the age of 21 years) diagnosed with a neoplastic disorder who have been offered NHSE whole genome sequencing.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — As per widely adopted clinical research practice for case reviews of de-identified, anonymised data, no explicit consent of participants (or their legal guardians) would be required for this study other than the consent they provided at biopsy (from which the whole genome sequencing data is derived) for researchers to access their notes (as documented on hospital consent form).

SUMMARY:
This retrospective case series reviews clinical notes to assess whether NHS whole genome sequencing provides tangible benefits for paediatric tumours.

DETAILED DESCRIPTION:
The NHSE-commissioned whole genome sequencing programme went live at the end of 2020. It remains as yet unproven, whether this whole genome sequencing programme for children with cancer can deliver tangible benefits in real-time. There is an urgent need, therefore, to assess whether children with tumours who are receiving NHS whole genome sequencing are actually benefiting from this additional assay. This is a retrospective case series. The principal methodology is that of reviewing clinical notes to assess whether children with tumours have benefited from NHSE whole genome sequencing. Apart from the contribution of our work to the scientific literature, this research will inform government on the potential benefits, or lack thereof, of the live NHSE whole genome programme and has the potential to influence policy on whether this programme should be continued.

ELIGIBILITY:
Inclusion Criteria:

* All children and young people (up to the age of 21 years) diagnosed with a neoplastic disorder who have been offered NHSE whole genome sequencing.

Exclusion Criteria:

* Anyone not offered NHSE whole genome sequencing
* Individuals beyond the age of 21
* Individuals without a neoplastic disorder.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children and young people (up to the age of 21 years) diagnosed with a neoplastic disorder
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of children clinically benefiting from whole genome sequencing | 5.5 years
  The proportion of children clinically benefiting from whole genome sequencing in terms of improving diagnoses, treatment, and prognostication, amongst other aspects

SECONDARY OUTCOMES:
Relation between mutation data and disease phenotypes | 5.5 years
  To describe possible associations between genetic features and clinical phenotypes. What these associations look like will depend on the study results.

OTHER OUTCOMES:
The cost of whole genome sequencing | 5.5 years
  The cost of whole genome sequencing versus standard of care assays as performed for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Wellcome Sanger Institute, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided